CLINICAL TRIAL: NCT02024750
Title: Family-Centered Tailoring of Pediatric Diabetes Self-Management Resources
Brief Title: Tailored Diabetes Self-Management Resources
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Medical College of Wisconsin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013-1506; MSN164403 (Other: Patient-Centered Outcomes Research Institute); IRB 00016300 (Other: Study Team)
Record Dates: First submitted 2013-12-27; First posted 2013-12-31 (Estimated); Results first posted 2019-09-18 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Family centered care; Patient centered care; Diabetes Mellitus, Type 1; Problem Recognition in Illness Self-Management (PRISM)
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tailored Resources (Experimental): Use of PRISM screening tool to identify self-management needs and to provide tailored group session resources over 1 year
  Interventions: Behavioral: Tailored Resources
- Usual Care (No Intervention): Patients and families obtain routine multidisciplinary diabetes care

INTERVENTIONS:
Behavioral: Tailored Resources — Based upon PRISM screening tool results that identifies self-management barriers, patient/family will receive self-management resources matched to their barriers. These resources could be focused on: 1. Understanding and organizing care; 2. Motivation to self-manage; and 3. Family Teamwork. Group session of about 6 families with the same barrier will meet four times fo 75-minutes over a year, at the clinic site on same date as routine clinic visit.
  Arms: Tailored Resources

SUMMARY:
Children with type 1 diabetes face complex self-management regimens which make adherence challenging and ultimately result in poor blood sugar control. Several common barriers interfere with diabetes control such as limited knowledge or challenges with staying motivated. Efficacious strategies exist to improve diabetes self-management including, but not limited to, diabetes education or family therapy. Patients and families often do not access these strategies, in part due to healthcare systems-based issues such as accessibility, provider availability, or insurance coverage.

A family-centered approach has been suggested to tailor diabetes care to provide improved outcomes for each child. Family-centered care engages the family in the decision-making about the child's health and well-being. In this study we will take a family-centered approach to providing diabetes self-management by identifying families' unique self-management barriers through a 10-minute survey tool called PRISM (Problem Recognition in Illness Self-Management). Based upon the results of PRISM, we will provide tailored self-management resources (interventions) to meet the family's needs. We will coordinate group-based delivery of the resources with routine diabetes clinic visits. These group-based resources will be delivered in four 75-minute sessions over a year.

The primary goal of this study is to compare the effectiveness of family-centered tailoring of diabetes self-management resources with the untailored approach of usual care. We hypothesize that the family-centered model of care with tailored resources will improve the outcomes of glycemic control and quality of life among children with type 1 diabetes and their parents.

DETAILED DESCRIPTION:
This project's long-term goal is to develop a system-level method to move existing, efficacious self-management resources into the hands of children with type 1 diabetes and their families. Over 175,000 US children have type 1 diabetes and face a lifetime of self-management decisions in an attempt to delay or prevent complications, avoid hypoglycemia, and maintain quality of life for themselves and their parents. Although efficacious self-management resources exist, most children with diabetes struggle to manage their disease. Several barriers to diabetes management exist, including knowledge, motivation, and family interactions. Because barriers are unique for each child and family, family-centered approaches are recommended. Currently, no systematic approach exists to identify and address each family's self-management barriers. Information from PRISM (Problem Recognition in Illness Self-Management), a 10-minute survey tool, could help families and clinicians make better decisions to address these barriers, ultimately improving outcomes, fostering family-centered diabetes care, and optimizing resource use.

This randomized, pragmatic trial will compare outcomes from PRISM-based, family-centered tailoring of self-management resources (intervention) to outcomes from the untailored approach of usual care. Our specific aims are to assess the effect of family-centered tailoring of diabetes self-management resources on outcomes that matter to the children and parents: glycemic control (A1c and fear of hypoglycemia) and child and parent quality of life.

Children 8-16 years old with diabetes (150 each in usual care and intervention groups) and their parents will be enrolled at two large pediatric diabetes clinics. We will 1) use PRISM to identify families' unique self-management barriers; 2) tailor self-management resources to identified barriers; and 3) coordinate group-based delivery of the resources with routine diabetes visits. The group-based resources will be delivered in four 75-minute sessions over 12 months. A1c will be assessed after sessions, along with fear of hypoglycemia and quality of life for the child and parent. We will compare outcomes with mixed-effects models.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents with type 1 diabetes and their parents who receive care at one of two sites in Wisconsin.
* Planning to continue care at clinic for the next 2 years.
* English speaking
* Diagnosed with diabetes for > 12 months

Exclusion Criteria:

* Newly diagnosed with diabetes (< 12 months)
* Participant in prior preliminary work for this study

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 214 (Actual)
Dates: Start 2014-09; Primary Completion 2017-08-08 (Actual); Study Completion 2017-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth D Cox, MD,PhD, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - University of Wisconsin - Madison, Madison, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fiallo-Scharer R, Palta M, Chewning BA, Rajamanickam V, Wysocki T, Wetterneck TB, Cox ED. Impact of family-centered tailoring of pediatric diabetes self-management resources. Pediatr Diabetes. 2019 Nov;20(7):1016-1024. doi: 10.1111/pedi.12899. Epub 2019 Aug 8. PMID 31355957
- [Derived] Fiallo-Scharer R, Palta M, Chewning BA, Wysocki T, Wetterneck TB, Cox ED. Design and baseline data from a PCORI-funded randomized controlled trial of family-centered tailoring of diabetes self-management resources. Contemp Clin Trials. 2017 Jul;58:58-65. doi: 10.1016/j.cct.2017.04.007. Epub 2017 Apr 24. PMID 28450194

RESULTS

PARTICIPANT FLOW:
Groups:
- Tailored Resources: Four 75-minute group-based self-management resource sessions, matched to self-management barriers identified by PRISM survey
- Usual Care: Routine multidisciplinary diabetes care
Period: Overall Study
Arm/Group | Tailored Resources | Usual Care
Started | 106 | 108
Completed | 104 | 107
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tailored Resources | Usual Care | Total
Number analyzed (Participants) | 106 | 108 | 214
Age, Customized [Count of Participants; unit: Participants]
  8-12 years old | 47 | 48 | 95
  13-16 years old | 59 | 60 | 119
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 59 | 105
  Male | 60 | 49 | 109
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Non-Hispanic, White | 87 | 92 | 179
  Race/Ethnicity: Not non-Hispanic, White | 18 | 16 | 34
  Race/Ethnicity: Unknown | 1 | 0 | 1
Clinical Site [Count of Participants; unit: Participants]
  Site 1 | 49 | 52 | 101
  Site 2 | 57 | 56 | 113
Relationship to child: Mother [Count of Participants; unit: Participants] | 84 | 97 | 181
Insulin pump use [Count of Participants; unit: Participants] | 62 | 48 | 110
Baseline A1c [Mean (Standard Deviation); unit: Percent A1c] | 8.9 (1.5) | 9.3 (1.7) | 9.1 (1.6)
Baseline Child Quality of Life (QOL) [Mean (Standard Deviation); unit: units on a scale] — Measured with PedsQL Diabetes Module, with values ranging 0-100 and higher values representing higher quality of life.
  units on a scale | 66.7 (13.7) | 66.0 (11.6) | 66.3 (12.7)
Baseline Parent Quality of Life (QOL) [Mean (Standard Deviation); unit: units on a scale] — Measured with PedsQL Family Impact Module, with values ranging 0-100 and higher values representing higher quality of life.
  units on a scale | 62.1 (15.1) | 60.4 (16.5) | 61.2 (15.8)
Baseline Parent Fear of Hypoglycemia (FOH) [Mean (Standard Deviation); unit: units on a scale] — Measured with the Worry Subscale from the Hypoglycemia Fear Survey Parent Version, with values ranging 0-75 and higher values representing greater fear of hypoglycemia.
  units on a scale | 38.0 (9.6) | 39.6 (10.3) | 38.8 (9.9)

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin A1c for Usual Care and Tailored Resources (Intervention) Arms, During and Post-Intervention
Description: Mean change in A1c per month (slope), during and post-intervention.
Time Frame: Up to 5 time points during the intervention (12 months) and up to 4 time points in the post-intervention period (12 months)
Population: 214 participants were analyzed for up to 5 time points during the intervention and up to 4 time points in the post-intervention period. Models include data to the point of withdrawal for 3 families.
Measure: Mean (Standard Error); unit: Percent HbA1c per month
Units Other Than Participants: HbA1c Observations
Groups:
- Usual Care: Participants who received usual care.
- Tailored Resources: Participants who received tailored resources.
Arm/Group | Usual Care | Tailored Resources
Number analyzed (Participants) | 108 | 106
Number analyzed (HbA1c Observations) | 784 | 798
Percent HbA1c per month
  During Intervention | 0.014 (0.009) | 0.018 (0.009)
  Post-Intervention | 0.035 (0.008) | 0.025 (0.008)
Statistical Analysis 1: Comparison: Usual Care vs Tailored Resources; During the intervention period, the treatment effect on A1c. Results reflect the difference in A1c trend between usual care and intervention arms; Test type: Other; p = 0.72, Mixed Models Analysis — The a priori threshold for statistical significance was p<0.05; Adjustments were made for study stratification variables and covariates that were imbalanced between study arms at baseline; Mean Difference (Net) = 0.005, 95% CI 2-sided [-0.021 to 0.030] — Negative values indicate a clinical benefit
Statistical Analysis 2: Comparison: Usual Care vs Tailored Resources; During the post-intervention period, the treatment effect on A1c. Results reflect the difference in A1c trend between usual care and intervention arms; Test type: Other; p = 0.38, Mixed Models Analysis — The a priori threshold for statistical significance was p<0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.010, 95% CI 2-sided [-0.034 to 0.013] — Negative values indicate a clinical benefit

2. Primary Outcome: Change in Child Quality of Life (QOL) for Usual Care and Tailored Resources (Intervention) Arms, During and Post-Intervention
Description: Mean change in child quality of life per month (slope), during and post-intervention. Child quality of life is measured by the PedsQL Diabetes Module. Possible scores range from 0 to 100 with higher scores indicating better quality of life. Positive slopes reflect improving quality of life.
Time Frame: Up to 2 time points during the intervention (12 months) and up to 3 time points in the post-intervention period (12 months)
Population: 214 participants were analyzed for up to 2 time points during the intervention and up to 3 time points in the post-intervention period. Models include data to the point of withdrawal for 3 families.
Measure: Mean (Standard Error); unit: QOL scores per month
Units Other Than Participants: Quality of Life Measures
Arm/Group | Usual Care | Tailored Resources
Number analyzed (Participants) | 108 | 106
Number analyzed (Quality of Life Measures) | 481 | 470
QOL scores per month
  During Intervention | 0.194 (0.096) | 0.217 (0.100)
  Post-Intervention | 0.083 (0.155) | 0.010 (0.163)
Statistical Analysis 1: Comparison: Usual Care vs Tailored Resources; During the intervention period, the treatment effect on child quality of life. Results reflect the difference in QOL trend between usual care and intervention arms; Test type: Other; p = 0.87, Mixed Models Analysis — The a priori threshold for statistical significance was p<0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.023, 95% CI 2-sided [-0.249 to 0.295] — Positive values indicate a clinical benefit
Statistical Analysis 2: Comparison: Usual Care vs Tailored Resources; During the post-intervention period, the treatment effect on child quality of life. Results reflect the difference in QOL trend between usual care and intervention arms; Test type: Other; p = 0.74, Mixed Models Analysis — The a priori threshold for statistical significance was p<0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.074, 95% CI 2-sided [-0.517 to 0.369] — Positive values indicate a clinical benefit

3. Primary Outcome: Change in Parent Quality of Life (QOL) for Usual Care and Tailored Resources (Intervention) Arms, During and Post-Intervention
Description: Mean change in parent quality of life per month (slope), during and post-intervention. Parent quality of life is measured by the PedsQL Family Impact Module. Possible scores range from 0 to 100 with higher scores indicating better quality of life. Positive slopes reflect improving quality of life.
Time Frame: as for outcome 2
Population: 214 parents were analyzed for up to 2 time points during the intervention and up to 3 time points in the post-intervention period. Models include data to the point of withdrawal for 3 families.
Measure: Mean (Standard Error); unit: QOL scores per month
Units Other Than Participants: Quality of Life Measures
Arm/Group | Usual Care | Tailored Resources
Number analyzed (Participants) | 108 | 106
Number analyzed (Quality of Life Measures) | 480 | 478
QOL scores per month
  During Intervention | 0.115 (0.097) | 0.078 (0.100)
  Post-Intervention | 0.182 (0.161) | 0.172 (0.168)
Statistical Analysis 1: Comparison: Usual Care vs Tailored Resources; During the intervention period, the treatment effect on parent quality of life. Results reflect the difference in QOL trend between usual care and intervention arms; Test type: Other; p = 0.79, Mixed Models Analysis — The a priori threshold for statistical significance was p<0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.037, 95% CI 2-sided [-0.312 to 0.237] — Positive values indicate a clinical benefit
Statistical Analysis 2: Comparison: Usual Care vs Tailored Resources; During the post-intervention period, the treatment effect on parent quality of life. Results reflect the difference in QOL trend between usual care and intervention arms; Test type: Other; p = 0.97, Mixed Models Analysis — The a priori threshold for statistical significance was p<0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.009, 95% CI 2-sided [-0.467 to 0.448] — Positive values indicate a clinical benefit

4. Secondary Outcome: Change In Parent Fear of Hypoglycemia (FOH) for Usual Care and Tailored Resources (Intervention) Arms, During and Post-Intervention
Description: Mean change in parent fear of hypoglycemia per month (slope), during and post-intervention. Parent fear of hypoglycemia is measured by the Hypoglycemia Fear Survey Worry Subscale. Possible scores range from 15 to 75 with higher scores indicating greater fear of hypoglycemia. Positive slopes reflect increasing fear of hypoglycemia.
Time Frame: Up to 2 time points during the intervention (12 months) and up to 2 time points in the post-intervention period (12 months)
Population: 214 parents were analyzed for up to 2 time points during the intervention and up to 2 time points in the post-intervention period. Models include data to the point of withdrawal for 3 families.
Measure: Mean (Standard Error); unit: FOH scores per month
Units Other Than Participants: Fear of Hypoglycemia Measures
Arm/Group | Usual Care | Tailored Resources
Number analyzed (Participants) | 108 | 106
Number analyzed (Fear of Hypoglycemia Measures) | 400 | 393
FOH scores per month
  During Intervention | -0.088 (0.089) | 0.046 (0.093)
  Post-Intervention | -0.074 (0.132) | -0.080 (0.139)
Statistical Analysis 1: Comparison: Usual Care vs Tailored Resources; During the intervention period, the treatment effect on parent fear of hypoglycemia. Results reflect the difference in FOH trend between usual care and intervention arms; Test type: Other; p = 0.30, Mixed Models Analysis — The a priori threshold for statistical significance was p<0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.134, 95% CI 2-sided [-0.121 to 0.388] — Positive values indicate a clinical benefit
Statistical Analysis 2: Comparison: Usual Care vs Tailored Resources; During the post-intervention period, the treatment effect on parent fear of hypoglycemia. Results reflect the difference in FOH trend between usual care and intervention arms; Test type: Other; p = 0.98, Mixed Models Analysis — The a priori threshold for statistical significance was p<0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.006, 95% CI 2-sided [-0.384 to 0.373] — Positive values indicate a clinical benefit

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Tailored Resources | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/106 | 0/108
Serious Adverse Events (participants affected / at risk) | 0/106 | 0/108
Other Adverse Events (participants affected / at risk) | 0/106 | 0/108

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-11-22): https://cdn.clinicaltrials.gov/large-docs/50/NCT02024750/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-22): https://cdn.clinicaltrials.gov/large-docs/50/NCT02024750/SAP_001.pdf